CLINICAL TRIAL: NCT07309198
Title: Effects and Mechanisms of Non-invasive Deep Brain Stimulation in Patients With Parkinson's Disease
Brief Title: Temporal Interference Stimulation on Motor Symptoms in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai University of Sport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 102772024RT146
Record Dates: First submitted 2025-11-15; First posted 2025-12-30 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease
Keywords: transcranial temporal interference stimulation; TIS; Parkinson's disease; motor symptoms
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIS Group (Experimental): Participants in this arm will receive active transcranial temporal interference stimulation targeting the internal globus pallidus over a two-week intervention period.
  Interventions: Device: Transcranial Temporal Interference Stimulation (TIS)
- Sham Group (Sham Comparator): Participants in this arm will receive sham transcranial temporal interference stimulation using the same electrode placement and experimental setup as the active intervention. The sham procedure consists of 10 sessions delivered over a two-week period, without therapeutic stimulation.
  Interventions: Device: Transcranial Temporal Interference Stimulation (TIS)

INTERVENTIONS:
Device: Transcranial Temporal Interference Stimulation (TIS) — Transcranial temporal interference stimulation (TIS) is a noninvasive brain stimulation technique that delivers two high-frequency alternating currents through scalp electrodes to generate a low-frequency interference field in deep brain regions. In this study, TIS targets the internal globus pallidus (GPi) to modulate neural activity in people with Parkinson's disease. Participants receive 10 stimulation sessions over two weeks. The sham TIS condition uses the same setup but applies low-frequency currents without generating an interference pattern.

SUMMARY:
The goal of this clinical trial is to learn whether a type of brain stimulation called transcranial temporal interference stimulation (TIS) of the internal globus pallidus (GPi) can help improve movement symptoms in people with Parkinson's disease. The study will also look at how TIS changes brain activity related to these improvements.

The main questions this study aims to answer are:

* How much can repeated TIS sessions improve movement symptoms in people with Parkinson's disease?
* Can these improvements last for up to two months after the treatment ends?
* What changes in brain activity happen along with the improvements?

Researchers will compare people who receive active TIS with those who receive sham (placebo-like) stimulation to see whether active TIS leads to better movement outcomes.

Participants will:

* Receive 10 sessions of active or sham TIS over two weeks
* Complete movement assessments during the two-week treatment and again 2, 4, and 8 weeks afterward
* Complete brain activity assessments before and after the two-week treatment

ELIGIBILITY:
Inclusion Criteria:

* A physician-diagnosed idiopathic Parkinson's disease (PD) according to the Movement Disorder Society (MDS) diagnostic criteria, with onset after the age of 40.
* Stable antiparkinsonian medication regimen, including levodopa-containing therapy, unchanged for at least 4 weeks before and during the trial.
* Hoehn and Yahr (H&Y) stages 1.5 to 3 and ability to walk unassisted.
* Absence of dementia, defined as a Montreal Cognitive Assessment (MoCA) score ≥ 21.

Exclusion Criteria:

* Any contraindication for MRI or transcranial temporal interference stimulation (TIS), including claustrophobia, metallic implants in the head or heart, or a history of electroconvulsive therapy.
* Current use of antipsychotic, antidepressant, or other dopamine-modulating medications.
* Presence of orthopedic conditions that may interfere with motor assessments, such as osteoarthritis or recent orthopedic surgery (within the past 6 months).
* History of physician-diagnosed major psychiatric illness.
* Physician-diagnosed cardiovascular risks that could contraindicate exercise or study participation.
* Prior history of deep brain stimulation (DBS) surgery.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
the Movement Disorder Society-Unified Parkinson's Disease Rating Scale-III (MDS-UPDRS III) Score | Baseline, immediately after 1 and 2 weeks of intervention, 2 weeks, 4 weeks, and 8 weeks after intervention.
  Change in motor symptoms assessed using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale-III (MDS-UPDRS III). The total score ranges from 0 to 132, with higher scores indicating more severe motor impairment (worse outcome).

SECONDARY OUTCOMES:
Home Diary Assessment of Motor States | Baseline, immediately after 1 and 2 weeks of intervention
  The motor state will be recorded by participants using a self-completed home diary during waking hours in 30-minute intervals from awakening until bedtime. For each interval, participants will record one of the following motor states: ON with good motor control, ON with mild dyskinesia, ON with severe dyskinesia, or OFF.
  Baseline assessment will be defined as the average percentage of waking time spent in ON states over three consecutive days immediately prior to the intervention. The 1-week assessment will be defined as the average percentage of waking time spent in ON states over the five intervention days of the first intervention week, and the 2-week assessment as the average over the five intervention days of the second intervention week.
  The outcome measure is defined as the percentage of total recorded waking time spent in ON states, calculated from the home diary data. A higher percentage of time spent in ON states indicates milder motor symptoms and better motor control.
Parkinson's Disease Questionnaire-39 (PDQ-39) Score | Baseline, immediately after 1 and 2 weeks of intervention, 2 weeks, 4 weeks, and 8 weeks after intervention.
  Change in quality of life assessed using the Parkinson's Disease Questionnaire-39 (PDQ-39). The PDQ-39 consists of 39 items across 8 domains, with total scores ranging from 0 to 100, where higher scores indicate poorer health-related quality of life (worse outcome).
the Movement Disorder Society-Unified Parkinson's Disease Rating Scale-I (MDS-UPDRS I) Score | Baseline, immediately after 1 and 2 weeks of intervention, 2 weeks, 4 weeks, and 8 weeks after intervention.
  Change in non-motor symptoms assessed using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale-I (MDS-UPDRS I) (Non-Motor Experiences of Daily Living). The total score ranges from 0 to 52, with higher scores indicating more severe non-motor symptoms (worse outcome).
the Movement Disorder Society-Unified Parkinson's Disease Rating Scale-II (MDS-UPDRS II) Score | Baseline, immediately after 1 and 2 weeks of intervention, 2 weeks, 4 weeks, and 8 weeks after intervention.
  Change in motor symptoms affecting daily living assessed using the Movement Disorder Society-Unified Parkinson's Disease Rating Scale-II (MDS-UPDRS II) (Motor Experiences of Daily Living). The total score ranges from 0 to 52, with higher scores indicating more severe motor difficulties in daily living (worse outcome).
Epworth Sleepiness Scale Score | Baseline, immediately after 1 and 2 weeks of intervention, 2 weeks, 4 weeks, and 8 weeks after intervention.
  Change in daytime sleepiness assessed using the Epworth Sleepiness Scale . The Epworth Sleepiness Scale is a self-administered questionnaire consisting of 8 items, with total scores ranging from 0 to 24, where higher scores indicate greater daytime sleepiness (worse outcome).
Parkinson's Disease Sleep Scale-2 Score | Baseline, immediately after 1 and 2 weeks of intervention, 2 weeks, 4 weeks, and 8 weeks after intervention.
  Change in sleep disturbances assessed using the Parkinson's Disease Sleep Scale-2.
  The Parkinson's Disease Sleep Scale-2 is a patient-reported questionnaire consisting of 15 items, with total scores ranging from 0 to 60, where higher scores indicate more severe sleep disturbances (worse outcome).
Gait Performance Measures | Baseline, immediately after 1 and 2 weeks of intervention, 2 weeks, 4 weeks, and 8 weeks after intervention.
  Changes in gait performance will be assessed using an instrumented gait mat during single-task and dual-task walking conditions.
  Spatiotemporal gait parameters, including gait speed, step length, stride length, step width, cadence, and gait variability, will be collected during standardized walking trials.
  Improvements in gait performance are indicated by increased gait speed, longer step and stride length, and reduced gait variability under both single-task and dual-task conditions.
Balance Performance Measures | Baseline, immediately after 1 and 2 weeks of intervention, 2 weeks, 4 weeks, and 8 weeks after intervention.
  Changes in balance performance will be assessed using a force platform during standardized standing balance tasks.
  Center of pressure (COP) parameters, including COP path length, sway area, and sway velocity, will be derived from force platform recordings to quantify postural stability.
  Improved balance performance is indicated by reduced COP displacement, smaller sway area, and lower sway velocity.
Magnetic Resonance Imaging (MRI) Measures | Baseline and immediately after the intervention
  Changes in brain structure and/or function will be assessed using magnetic resonance imaging (MRI).
  MRI data will be acquired to evaluate intervention-related changes in brain regions associated with motor control. Imaging-derived measures may include structural and functional metrics obtained from standardized MRI protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai University of Sport, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No